CLINICAL TRIAL: NCT06001619
Title: Prostate Medication, Metabolism and Gut Microbiota
Acronym: PROMED
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-500618-24-00
Record Dates: First submitted 2023-04-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Prostatic Hyperplasia; Prostate Cancer
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Neoplasms | interventions — Finasteride; Dutasteride; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prostatic hyperplasia (Experimental): Inclusion criteria for the BPH cohort includes clinical decision to initiate treatment of benign prostate hyperplasia (BPH) with 5-alpha-reductase inhibitors (finasteride, dutasteride, or combination of dutasteride and tamsulosin). Before starting the medication, size of the prostate has been measured with TRUS (transrectal ultrasound). The BPH cohort will include a total of 50 subjects and the study samples (gut microbiota, metabolite sampling) will be collected prior the start of the 5-alpha- reductase inhibitors and after 2 months of medical therapy. At this stage, PSA is determined from blood sample and the size of the prostate is measured with transrectal ultrasound (TRUS). In addition, after 6 months, PSA and prostate size measurements are repeated.
  Interventions: Drug: Prostate hyperplasia medication
- Prostatic cancer (Experimental): Inclusion criteria for the cancer cohort include a clinical decision to initiate PCa treatment with androgen deprivation therapy (ADT) with LHRH antagonist (degarelix). This may include either treatment of a metastatic disease with definite ADT or adjuvant ADT to external beam radiation of the prostate. The cancer cohort will include a total of 50 subjects and the study samples (gut microbiota, metabolite sampling) will be collected prior the start of the ADT and after 2 months of medical therapy. In addition, after 2 and 6 months, PSA measurement is repeated.
  Interventions: Drug: LhRH-antagonist

INTERVENTIONS:
Drug: Prostate hyperplasia medication — The dosages prostatic hyperplasia medication: dutasteride 0,5 MG x1 or finasteride 5 MG x1 or combination of dutasteride and tamsulosin 0,5/0,4 MG x1.
  Other Names: Finasteride 5 MG; Dutasteride 0,5 MG; Dutasteride and Tamsulosin 0,5/0,4 MG
  Arms: Prostatic hyperplasia
Drug: LhRH-antagonist — The starting dose in prostatic cancer patient cohort of LHRH antagonist degarelix is 120 MGx2 and the maintenance dose is 80 MGx1.
  Other Names: Degarelix 120 MG
  Arms: Prostatic cancer

SUMMARY:
PROMED is a prospective, single center translational multiple cohort study to investigate the association of prostate medication and gut microbiota. The main aim is to investigate how prostate hormonal therapy (5-ARI, ADT) affects gut microbiota composition. Aalso study metabolic characteristics in the gut and systemic circulation in men with different medications will be studied. In addition, the effect of gut microbiota on patient's response to medications will be investigated. The medicines used in the study to treat benign prostate hyperplasia are dutasteride and finasteride and a combination of dutasteride and tamsulosin. LHRH antagonist degarelix is used as a medication to treat patients with cancer. The dosages of 5-ARI medication: dutasteride 0,5mg x1 or finasteride 5mg x1 or combination of dutasteride and tamsulosin 0,5/0,4mg x1. The starting dose of LHRH antagonist degarelix is 120mgx2 and the maintenance dose is 80mgx1. The medication for PCa is planned according to the protocol but so that each subject receives degarelix at the beginning of treatment and one month after initiation. Thereafter, the medication is continued according to the clinician's assessment. The study is carried out in Turku University Hospital and University of Turku.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is a significant health care system challenge. PCa is the most common male cancer in Finland and most western countries. Interestingly, although the incidence of indolent (latent) PCa is very similar throughout the globe, there is a remarkable global age-adjusted incidence variation (up to 40-fold difference between highest and lowest incidences).

Epidemiological data suggest that aging in men is associated with neoplastic processes in the prostate but only a subset of men will develop a true malignancy potentially affecting their life-span or quality of life. Genetic factors have a significant effect on PCa risk, but very likely life-style (e.g. diet and physical activity) affect PCa risk as well, but the mechanisms mediating protective or harmful effects of life-style remain unclear.

Gut microbiota, i.e. the collection of microbes colonizing the gastrointestinal tract, is acknowledged to play significant role in many metabolic pathways and pathogenic processes in the human body. Although there is some evidence suggesting that gut microbiota affects therapy responses (especially androgen deprivation) in PCa, it ́s potential role in prostate carcinogenesis is not well documented. Our previous studies suggest that gut microbiota composition is different in men with and without PCa and that changes in steroid hormone synthesis may be one mechanism how gut microbiota affects PCa risk.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Ability and stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* Any history of a fecal transplantation.
* Recent (within 3 months or still symptomatic) gastroenteritis.
* Antibiotic treatment within 3 months (expect for antibiotic prophylaxis related to prostate biopsies).
* Inability to comply with the protocol of unwillingness to participate in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostatic diseases
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota signature before 5-ARI therapy | before starting prostate 5-ARI medication
  Gut microbiota signature before 5-ARI therapy
Gut microbiota signature after 5-ARI therapy | 2 months after starting prostate 5-ARI medication
  Gut microbiota signature after 5-ARI therapy
Gut microbiota signature before ADT (LHRH antagonists). | before starting prostate degarelix
  Gut microbiota signature before ADT (LHRH antagonists).
Gut microbiota signature after ADT (LHRH antagonists). | 2 months after starting prostate degarelix
  Gut microbiota signature after ADT (LHRH antagonists).

SECONDARY OUTCOMES:
Metabolic characteristics in the gut and systemic circulation after use of prostate medication | before starting prostate idcation (degarelix or finasteride/dutasteride)
  Gut metabolic charachteristics of men receiving prostate medication
Metabolic characteristics in the gut and systemic circulation before iuse of prostate medication | 2 months after from starting prostate medication (degarelix or finasteride/d
  Gut metabolic charachteristics of men receiving prostate medication

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Turku University Hospital, Turku
  - University of Turku, Turku